CLINICAL TRIAL: NCT05958225
Title: SEE Change Evaluation - Assessing Impacts of Personal Agency Training to Advance Entrepreneurial Outcomes in Uganda
Brief Title: SEE Change Evaluation - Impacts of Personal Agency Training on Ugandan Entrepreneurs
Acronym: SEE-Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Investors Club/Enterprise Uganda (Unknown); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024029
Record Dates: First submitted 2023-06-26; First posted 2023-07-24 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Well-Being, Psychological; Economic Hardship; Stress
Keywords: Personal agency; entrepreneurship; flourishing
MeSH Terms: conditions — Psychological Well-Being; Financial Stress

STUDY DESIGN:
Intervention Model Description: Participants will be randomly selected (using a stratified random sampling, stratified by gender) and assigned to either the intervention group (n=400) or wait-listed control group (n=400).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal agency, leadership and business training (Experimental): Entrepreneurs will participate in a 3 day residential training (based on SEE Change's Empowered Entrepreneur training) that integrates personal agency with basic business and leadership topics. Participants will also get weekly support messages on their phone for 6 weeks and a check in by a training once a month for 3 months.
  Interventions: Behavioral: SEE Change Business and Personal Agency Training
- Control (No Intervention): For this study, the control participants will not receive any intervention.

INTERVENTIONS:
Behavioral: SEE Change Business and Personal Agency Training — A three day residential training based on SEE Change's Empowered Entrepreneur Training curriculum. This training will be led by a certified SEE Change trained facilitator. The workshop will include individual and group exercises that allow participants to increase their self-awareness, build mental tools for resiliency and adaptability in their life, create life visions and key tools to create behavior change. Additional exercises will include specific business related content including record keeping, financial planning and marketing strategies based on the Business Model Canvas tool.
  After the 3 day training, the participants will receive a supportive message through an interactive voice recording, once a week for 6 weeks. In addition, they will be contacted once a month, for three months (either by phone or in person) by the trainer to see how they are doing on their goals.
  Arms: Personal agency, leadership and business training

SUMMARY:
This study is proposed as an individually randomized control trial (RCT) designed to assess the short-term impacts (follow up at six months) of a personal agency training on a range of economic and health outcomes for micro and small entrepreneurs in Western and Central Uganda. Participants will be randomly selected and assigned to either the intervention group (n=400) or wait-listed control group (n=400). The intervention will include the standard Empowered Entrepreneur training curriculum which includes personal agency alongside basic business training that has been developed by the SEE Change team. This training will take place over three consecutive days (approximately 25 hours of content).

DETAILED DESCRIPTION:
The investigators propose to examine the comparative impacts of a personal agency and business training curricula on outcome measures focused in three areas 1) business related outcomes; 2) personal agency and flourishing; and 3) social spillover impacts.

Aim 1: Assess changes in business related outcomes including improved sales and profit, enhanced business skills and behaviors, and business-related goal setting.

Aim 2: Assess changes in personal agency and flourishing as determined through personal goal setting and psychometric measurements of self-esteem, self-confidence, grit and flourishing.

Aim 3: Assess social spillover impacts of the training on depression, anxiety and stress, and changes in gender norms and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Small or micro entrepreneur;
* Business has been in operation/existence for at least the past 12 months;
* Entrepreneur is between the ages of 18 and 55;
* Entrepreneur has the ability to participate in all training activities;
* Informed consent is obtained from the entrepreneur;
* The entrepreneur is not planning to leave the area in the next 12 months;
* The entrepreneur has access to a phone for contact purposes;

Exclusion Criteria:

* Entrepreneur is unable to provide informed consent or informed consent is not obtained;
* Entrepreneur is not considered a small or micro entrepreneur;
* Entrepreneur is younger than 18 years of age;
* Business has been in operation/existence for less than 12 months;
* Entrepreneur's primary business is farming (anything related to seasonal crop production);
* Entrepreneur is planning to leave the area in the next 12 months;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 814 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Business revenue and profits as assessed by questionnaire developed by study team | Baseline, six months
  Specific questions to assess types of income generating activities and overall business growth over the past month. Questions include number of income generating activities, length of time in business, business type, days and hours worked in business, number of employees, revenues and profits earned in business. Each of these questions can be examined separately or together as a composite score based on the number of questions are combined together.
Change in Marketing score as assessed by questionnaire as assessed by the Micro-Enterprise survey | Baseline, six months
  A composite score made up of a list of marketing activities that have been completed over the past three months. The score range is 0-10, with 0 being the lowest marketing activities to 10 as using all of the marketing strategies mentioned. There are 10 activities asked about (as yes/no questions) include questions to assess: negotiating with suppliers, engaging with customers to learn their needs or provide special offers, keeping supplies stocked and visiting competitors businesses.
Change in in the number of Marketing strategies adopted as assessed by questionnaire developed by study team | Baseline, six months
  A composite score made up of a list of types of marketing strategies that have been completed over the past six months. The score is assess from 0-8 and includes affirmative responses. Having a score of 0 is lowest, and 8 is the highest level of marketing strategies
Change in adoption of Business skills as assessed by questionnaire developed by study team | Baseline, six months
  A composite score made up of responses to a list of key business skills utilized over the past six months. These 10 questions include topics such as record keeping, keeping balance sheets, financial planning, understanding which items lead to higher profits, analysis of financial performance. Having a score of 0 is lowest, and 10 is the highest in terms of business skills.
Change in Self-efficacy as measured by the Chen scale for self efficacy | Baseline, six months
  This scale asks 8 questions related to self-efficacy and each question is scored on a likert scale from 1 (Strongly disagree) to 5 (Strongly agree). The range of score are from 8-40, but usually examined as an average score (1-5), with the lowest scores being very low self-efficacy and the highest score being high self-efficacy.
Change in Self-esteem as measured by the Rosenberg scale | Baseline, six months
  The Self-esteem scale is a 10 question scales that is scored on a Likert scale of 1 (strongly disagree) to 5 (strongly agree). The total score range is 10-50 and is usually examined as an average score (1-5), with the lowest scores indicating very low self-esteem and the highest score indicating very high self-esteem
Change in ability to regulate behavior as assessed by the Short Self-Regulation Questionnaire (SSRQ) | Baseline, six months
  The Short Self-Regulation Questionnaire (SSRQ) is a 31-item measure of the ability to regulate behavior in order to achieve desired future outcomes. Each question is scored on a Likert scale of 1 (strongly disagree) to 5 (strongly agree), with the lowest score indicating low level of self-regulation to the highest level of self-regulation - with a range of 31-155 after adjustments for reverse scoring

SECONDARY OUTCOMES:
Change in perseverance assessed by the Grit scale | Baseline, six months
  The Grit scales includes 10 questions designed to assess level of perseverance, ability to overcome challenges and move towards one's goals. Each question is score on a Likert scale of 1 (strongly disagree) to 5 (strongly agree), with the lowest scores indicating very low grit and the highest scores indicating very high levels of grit, range (10-50)
Change in Locus of control as measured by the Internal-External Locus of Control Short Scale-4 (IE-4) | Baseline, six months
  This short scale consists of 4 questions to assess how much individuals feel that have control over their lives. These questions are scored on a Likert scale from 1 (strongly disagree) to 5 (strongly agree) with the lowest scores (2) for the first two questions indicating that the individuals has a low sense of internal control over their lives, but if they score high on the first two questions (10), it indicates a high level of internal control. Similarly low scores on the remaining 2 questions indicate a low level of external control and high scores indicate a high level of external control on their lives.
Change in understanding of gender norms as assessed by the Gender norms and attitude scale | Baseline, six months
  This 14 question scales is focused on understanding gender norms of the participant. Each question is scored via a Likert scale from 1 (strongly agree) to 5 (strongly disagree). Some of the questions are reverse scored, however, the scale is averaged to scores of 1-5 with the lowest scores indicating beliefs that are more in line with traditional gender norms and high scores indicating beliefs for greater equity for women, with a range of 14-70 or an average score 1-5.
Change in Depression Anxiety and Stress Scale (DASS 8) | Baseline, six months
  This 8 question psychometric scale is a shortened version of the DASS 21 scale and covers questions referring to symptoms of depression, anxiety and stress. Participants are asked to rate whether they strongly agree or strongly disagree on a 6 point scale. The first 4 questions are focused on depression with a scale range of 4-24 and questions 5-8 are focused on anxiety (with a similar scale range). The lowest scores correspond to better outcomes related to depression or anxiety and the highest score correspond to worse levels of depression or anxiety.
Change in environmental mastery as assessed by the Ryff Environmental Mastery subscale | Baseline, six months
  The environmental mastery scale is a subscale of the larger Ryff scales for social agency. It has 9 questions that are scored via a Likert scale of 1 (strongly disagree) and 5 (strongly agree). Some of the questions are reverse scored, but the final scores relate to high levels (5) or low levels (1) of environmental mastery.
Change in positive relations as assessed by the Ryff Positive Relations with Others subscale | Baseline, six months
  The positive relations with others scale is a subscale of the larger Ryff scales for social agency. It has 9 questions that are scored via a Likert scale of 1 (strongly disagree) and 5 (strongly agree). Some of the questions are reverse scored, but the final scores relate to high levels (5) or low levels (1) of positive relationships with others.
Change in personal initiative as assessed by the Personal Initiative Scale | Baseline, six months
  This 9 question scale was developed to assess level of personal initiative, drawing from their personal agency. This scales helps examine an individual's ability to be proactive and each question is scored via a Likert scale from 1 (strongly disagree) to 5 (strongly agree). An aggregate score is developed with the lowest scores indicating a low level of personal initiative and a high score as having a high level of personal initiative.

CONTACTS AND LOCATIONS:
Overall Officials: Anita V Shankar, PhD, Principal Investigator — Associate Scientist, Johns Hopkins School of Public Health
Locations (1):
- Innovations for Poverty Action, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Mel, Suresh and McKenzie, David John and Woodruff, Christopher, Business Training and Female Enterprise Start-Up, Growth, and Dynamics: Experimental Evidence from Sri Lanka (July 1, 2012). World Bank Policy Research Working Paper No. 6145
- [Background] Chen, G., Gully, S. M., & Eden, D. (2001). Validation of a new general self-efficacy scale. Organizational research methods, 4(1), 62-83.
- [Background] Duckworth AL, Quinn PD. Development and validation of the short grit scale (grit-s). J Pers Assess. 2009 Mar;91(2):166-74. doi: 10.1080/00223890802634290. PMID 19205937
- [Background] Robins, R. W., Hendin, H. M., & Trzesniewski, K. H. (2001). Measuring global self-esteem: Construct validation of a single-item measure and the Rosenberg Self-Esteem Scale. Personality and social psychology bulletin, 27(2), 151-161.
- [Background] Rosenberg, M. (1965). Rosenberg self-esteem scale (RSE). Acceptance and commitment therapy. Measures package, 61(52), 18.
- [Background] Kovaleva, A., Beierlein, C., Kemper, C. J., & Rammstedt, B. (2014). Internale-Externale-Kontrollüberzeugung-4 (IE-4). Zusammenstellung sozialwissenschaftlicher Items und Skalen (ZIS). https://doi.org/10.6102/zis184
- [Background] Niessen D, Schmidt I, Groskurth K, Rammstedt B, Lechner CM. The Internal-External Locus of Control Short Scale-4 (IE-4): A comprehensive validation of the English-language adaptation. PLoS One. 2022 Jul 11;17(7):e0271289. doi: 10.1371/journal.pone.0271289. eCollection 2022. PMID 35816496
- [Background] Waszak, C, JL Severy, L Kafafi, and I Badawi. 2000. Fertility behavior and psychological stress: The mediating influence of gender norm beliefs among Egyptian women. Psychology of Women Quarterly 25:197-208.
- [Background] VanderWeele TJ, McNeely E, Koh HK. Reimagining Health-Flourishing. JAMA. 2019 May 7;321(17):1667-1668. doi: 10.1001/jama.2019.3035. No abstract available. PMID 30933213
- [Background] Norton PJ. Depression Anxiety and Stress Scales (DASS-21): psychometric analysis across four racial groups. Anxiety Stress Coping. 2007 Sep;20(3):253-65. doi: 10.1080/10615800701309279. PMID 17999228
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Carey KB, Neal DJ, Collins SE. A psychometric analysis of the self-regulation questionnaire. Addict Behav. 2004 Feb;29(2):253-60. doi: 10.1016/j.addbeh.2003.08.001. PMID 14732414